CLINICAL TRIAL: NCT07314268
Title: ATTR Amyloid Cardiomyopathy: Characterization of Extracellular Vesicles as Potential Disease Stratifiers and Prognostic Biomarkers
Acronym: EV-ATTR
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, FELIX JOSÉ ALVAREZ RAMIRES, Principal Investigator, University of Sao Paulo General Hospital
Other Study IDs: 83160124.2.0000.0068
Record Dates: First submitted 2025-11-25; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Wild-type ATTR Amyloidosis; Amyloidosis Cardiac; Amyloidosis, Hereditary; Amyloidosis Transthyretin
Keywords: Early Diagnosis; Serum Biomarkers; Transthyretin Amyloid Cardiomyopathy; ATTR; Vesicle Protein Signature
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis, Familial; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Serum samples will be collected and processed for isolation of circulating extracellular vesicles. Aliquots will be stored for proteomic, molecular, and vesicle characterization analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- TTR-CA + DM: TTR amyloid cardiomyopathy and myocardial dysfunction
- TTR-A: TTR amyloidosis and neurological involvement
- TTR-Gen: TTR amyloid genotype without phenotypic expression
- CTL: healthy controls

SUMMARY:
This study explores whether extracellular vesicles (EVs) tiny particles released into the bloodstream by cells can serve as early and minimally invasive biomarkers for transthyretin amyloid cardiomyopathy (ATTR-CM). Because ATTR-CM is often diagnosed only after significant heart damage has occurred, there is an urgent need for earlier detection methods.

The study will enroll individuals with different clinical presentations of transthyretin amyloidosis, along with healthy controls. Participants will undergo blood sampling, cardiac imaging (including echocardiography, cardiac MRI, and scintigraphy when indicated), and molecular EV analysis.

By comparing EV profiles across groups, the study aims to determine whether these vesicles reflect early cardiac involvement, track disease progression, and support more accurate and timely diagnosis. Ultimately, this research seeks to improve clinical decision-making and patient outcomes in ATTR cardiomyopathy.

DETAILED DESCRIPTION:
Transthyretin amyloid cardiomyopathy (ATTR-CM) is a progressive infiltrative disease caused by the deposition of misfolded transthyretin protein in the myocardium. Despite advances in imaging and treatment, early detection and accurate risk stratification remain major challenges, often resulting in delayed diagnosis and worse clinical outcomes.

This prospective observational study will enroll 70 adult participants, distributed into four predefined groups:

* ATTR-CM with myocardial dysfunction (n = 20)
* Hereditary ATTR with predominant neurologic involvement (n = 20)
* Genotype-positive individuals without clinical manifestation (n = 10)
* Healthy controls (n = 20)

All participants will undergo blood collection for extracellular vesicle (EV) isolation and molecular profiling. EVs are nanoscale particles released by cells that carry proteins, lipids, and nucleic acids reflective of their cellular origin and physiological state, potentially serving as minimally invasive biomarkers.

Participants with cardiac involvement will additionally undergo standardized cardiac evaluations, including echocardiography, cardiac MRI, and nuclear imaging when indicated. Clinical data, functional status, and laboratory parameters will be correlated with EV characteristics to assess their association with disease severity and progression.

By integrating EV profiling with clinical and imaging findings across different phenotypes and disease stages, this study aims to identify biomarkers capable of improving diagnostic accuracy, tracking disease evolution, and supporting personalized care strategies in ATTR amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older;
* Confirmed diagnosis of transthyretin cardiac amyloidosis (TTR-CA), with or without myocardial dysfunction, according to established diagnostic criteria;
* Willingness to comply with study procedures and requirements;
* Ability to provide written informed consent.

Exclusion Criteria:

* Presence of other significant cardiac conditions that may interfere with study outcomes, such as severe coronary artery disease or major valvular disease;
* Inability to provide informed consent or to participate in the required clinical assessments and examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult participants aged 18 years or older, including patients with confirmed transthyretin cardiac amyloidosis (with or without myocardial dysfunction), as well as healthy volunteers without known cardiac disease. The population includes individuals with different clinical presentations of ATTR and matched controls for comparative analysis.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum concentration of circulating extracellular vesicles (EVs) | baseline
  Quantification of the total concentration of circulating extracellular vesicles isolated from peripheral blood, expressed as number of particles per mL, measured by Nanoparticle Tracking Analysis (NTA - NanoSight), in participants with different clinical presentations of transthyretin amyloidosis (ATTR) and in healthy controls.
Circulating extracellular vesicle protein profile | baseline
  Protein profiling of circulating extracellular vesicles isolated from peripheral blood, including protein identification and assessment of relative abundance by mass spectrometry, followed by targeted validation and quantification of selected proteins using Western blotting and/or ELISA. Results will be reported as relative protein expression intensity or, when applicable, as absolute concentration (ng/mL), in participants with transthyretin amyloidosis (ATTR) and healthy controls, assessed at baseline.

SECONDARY OUTCOMES:
Correlation between circulating extracellular vesicle concentration and echocardiographic parameters | baseline
  Correlation between plasma concentration of circulating extracellular vesicles, measured as particles/mL by Nanoparticle Tracking Analysis, and cardiac structure and function parameters assessed by transthoracic echocardiography, including interventricular septal thickness (mm), left ventricular ejection fraction (%), and global longitudinal strain (%), analyzed using Pearson or Spearman correlation coefficients as appropriate, in participants with transthyretin amyloidosis (ATTR) and healthy controls.
Correlation between extracellular vesicle molecular profile and cardiac magnetic resonance findings | baseline
  Correlation between the molecular profile of circulating extracellular vesicles, including protein levels assessed by Western blotting and/or ELISA and microRNA expression assessed by RT-qPCR, and cardiac involvement parameters evaluated by cardiac magnetic resonance imaging, including extracellular volume fraction (ECV, %) and presence or absence of late gadolinium enhancement, analyzed using correlation methods as appropriate, in participants with transthyretin amyloidosis (ATTR) and healthy controls.
Correlation between extracellular vesicle characteristics and myocardial uptake on scintigraphy | baseline
  Correlation between circulating extracellular vesicle concentration, measured as particles/mL by Nanoparticle Tracking Analysis, and extracellular vesicle molecular characteristics assessed by RT-qPCR and Western blotting, and the degree of myocardial uptake evaluated by bone scintigraphy using an appropriate radiotracer and visual scoring system (e.g., Perugini grade 0-3), analyzed using correlation methods as appropriate, in participants with transthyretin amyloidosis (ATTR) and healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coracao, HCFMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Perez-Gonzalez R, Kim Y, Miller C, Pacheco-Quinto J, Eckman EA, Levy E. Extracellular vesicles: where the amyloid precursor protein carboxyl-terminal fragments accumulate and amyloid-beta oligomerizes. FASEB J. 2020 Sep;34(9):12922-12931. doi: 10.1096/fj.202000823R. Epub 2020 Aug 9. PMID 32772431
- [Background] Moreno CR, Ramires JAF, Lotufo PA, Soeiro AM, Oliveira LMDS, Ikegami RN, Kawakami JT, Pereira JJ, Reis MM, Higuchi ML. Morphomolecular Characterization of Serum Nanovesicles From Microbiomes Differentiates Stable and Infarcted Atherosclerotic Patients. Front Cardiovasc Med. 2021 Aug 5;8:694851. doi: 10.3389/fcvm.2021.694851. eCollection 2021. PMID 34422924
- [Background] Roura S, Gamez-Valero A, Lupon J, Galvez-Monton C, Borras FE, Bayes-Genis A. Proteomic signature of circulating extracellular vesicles in dilated cardiomyopathy. Lab Invest. 2018 Oct;98(10):1291-1299. doi: 10.1038/s41374-018-0044-5. Epub 2018 Mar 14. PMID 29540862
- [Background] Bakhshandeh B, Kamaleddin MA, Aalishah K. A Comprehensive Review on Exosomes and Microvesicles as Epigenetic Factors. Curr Stem Cell Res Ther. 2017;12(1):31-36. doi: 10.2174/1574888x11666160709211528. PMID 27396390
- [Background] van der Pol E, Hoekstra AG, Sturk A, Otto C, van Leeuwen TG, Nieuwland R. Optical and non-optical methods for detection and characterization of microparticles and exosomes. J Thromb Haemost. 2010 Dec;8(12):2596-607. doi: 10.1111/j.1538-7836.2010.04074.x. PMID 20880256
- [Background] Ridger VC, Boulanger CM, Angelillo-Scherrer A, Badimon L, Blanc-Brude O, Bochaton-Piallat ML, Boilard E, Buzas EI, Caporali A, Dignat-George F, Evans PC, Lacroix R, Lutgens E, Ketelhuth DFJ, Nieuwland R, Toti F, Tunon J, Weber C, Hoefer IE. Microvesicles in vascular homeostasis and diseases. Position Paper of the European Society of Cardiology (ESC) Working Group on Atherosclerosis and Vascular Biology. Thromb Haemost. 2017 Jun 28;117(7):1296-1316. doi: 10.1160/TH16-12-0943. Epub 2017 Jun 1. PMID 28569921
- [Background] Sunkara V, Woo HK, Cho YK. Emerging techniques in the isolation and characterization of extracellular vesicles and their roles in cancer diagnostics and prognostics. Analyst. 2016 Jan 21;141(2):371-81. doi: 10.1039/c5an01775k. PMID 26535415
- [Background] Roy S, Hochberg FH, Jones PS. Extracellular vesicles: the growth as diagnostics and therapeutics; a survey. J Extracell Vesicles. 2018 Feb 26;7(1):1438720. doi: 10.1080/20013078.2018.1438720. eCollection 2018. PMID 29511461
- [Background] Stremersch S, De Smedt SC, Raemdonck K. Therapeutic and diagnostic applications of extracellular vesicles. J Control Release. 2016 Dec 28;244(Pt B):167-183. doi: 10.1016/j.jconrel.2016.07.054. Epub 2016 Aug 2. PMID 27491882
- [Background] Gillmore JD, Maurer MS, Falk RH, Merlini G, Damy T, Dispenzieri A, Wechalekar AD, Berk JL, Quarta CC, Grogan M, Lachmann HJ, Bokhari S, Castano A, Dorbala S, Johnson GB, Glaudemans AW, Rezk T, Fontana M, Palladini G, Milani P, Guidalotti PL, Flatman K, Lane T, Vonberg FW, Whelan CJ, Moon JC, Ruberg FL, Miller EJ, Hutt DF, Hazenberg BP, Rapezzi C, Hawkins PN. Nonbiopsy Diagnosis of Cardiac Transthyretin Amyloidosis. Circulation. 2016 Jun 14;133(24):2404-12. doi: 10.1161/CIRCULATIONAHA.116.021612. Epub 2016 Apr 22. PMID 27143678
- [Background] Fontana M, Pica S, Reant P, Abdel-Gadir A, Treibel TA, Banypersad SM, Maestrini V, Barcella W, Rosmini S, Bulluck H, Sayed RH, Patel K, Mamhood S, Bucciarelli-Ducci C, Whelan CJ, Herrey AS, Lachmann HJ, Wechalekar AD, Manisty CH, Schelbert EB, Kellman P, Gillmore JD, Hawkins PN, Moon JC. Prognostic Value of Late Gadolinium Enhancement Cardiovascular Magnetic Resonance in Cardiac Amyloidosis. Circulation. 2015 Oct 20;132(16):1570-9. doi: 10.1161/CIRCULATIONAHA.115.016567. Epub 2015 Sep 11. PMID 26362631
- [Background] Maurer MS, Elliott P, Comenzo R, Semigran M, Rapezzi C. Addressing Common Questions Encountered in the Diagnosis and Management of Cardiac Amyloidosis. Circulation. 2017 Apr 4;135(14):1357-1377. doi: 10.1161/CIRCULATIONAHA.116.024438. PMID 28373528
- [Background] Gonzalez-Lopez E, Gagliardi C, Dominguez F, Quarta CC, de Haro-Del Moral FJ, Milandri A, Salas C, Cinelli M, Cobo-Marcos M, Lorenzini M, Lara-Pezzi E, Foffi S, Alonso-Pulpon L, Rapezzi C, Garcia-Pavia P. Clinical characteristics of wild-type transthyretin cardiac amyloidosis: disproving myths. Eur Heart J. 2017 Jun 21;38(24):1895-1904. doi: 10.1093/eurheartj/ehx043. PMID 28329248
- [Background] Treibel TA, Fontana M, Gilbertson JA, Castelletti S, White SK, Scully PR, Roberts N, Hutt DF, Rowczenio DM, Whelan CJ, Ashworth MA, Gillmore JD, Hawkins PN, Moon JC. Occult Transthyretin Cardiac Amyloid in Severe Calcific Aortic Stenosis: Prevalence and Prognosis in Patients Undergoing Surgical Aortic Valve Replacement. Circ Cardiovasc Imaging. 2016 Aug;9(8):e005066. doi: 10.1161/CIRCIMAGING.116.005066. PMID 27511979
- [Background] Galat A, Guellich A, Bodez D, Slama M, Dijos M, Zeitoun DM, Milleron O, Attias D, Dubois-Rande JL, Mohty D, Audureau E, Teiger E, Rosso J, Monin JL, Damy T. Aortic stenosis and transthyretin cardiac amyloidosis: the chicken or the egg? Eur Heart J. 2016 Dec 14;37(47):3525-3531. doi: 10.1093/eurheartj/ehw033. Epub 2016 Feb 22. PMID 26908951
- [Background] Ruberg FL, Berk JL. Transthyretin (TTR) cardiac amyloidosis. Circulation. 2012 Sep 4;126(10):1286-300. doi: 10.1161/CIRCULATIONAHA.111.078915. No abstract available. PMID 22949539
- [Background] Mankad AK, Shah KB. Transthyretin Cardiac Amyloidosis. Curr Cardiol Rep. 2017 Aug 24;19(10):97. doi: 10.1007/s11886-017-0911-5. PMID 28840452
- [Background] Damy T, Costes B, Hagege AA, Donal E, Eicher JC, Slama M, Guellich A, Rappeneau S, Gueffet JP, Logeart D, Plante-Bordeneuve V, Bouvaist H, Huttin O, Mulak G, Dubois-Rande JL, Goossens M, Canoui-Poitrine F, Buxbaum JN. Prevalence and clinical phenotype of hereditary transthyretin amyloid cardiomyopathy in patients with increased left ventricular wall thickness. Eur Heart J. 2016 Jun 14;37(23):1826-34. doi: 10.1093/eurheartj/ehv583. Epub 2015 Nov 3. PMID 26537620
- [Background] Maleszewski JJ. Cardiac amyloidosis: pathology, nomenclature, and typing. Cardiovasc Pathol. 2015 Nov-Dec;24(6):343-50. doi: 10.1016/j.carpath.2015.07.008. Epub 2015 Aug 1. PMID 26361138
- [Background] Banypersad SM, Moon JC, Whelan C, Hawkins PN, Wechalekar AD. Updates in cardiac amyloidosis: a review. J Am Heart Assoc. 2012 Apr;1(2):e000364. doi: 10.1161/JAHA.111.000364. Epub 2012 Apr 24. No abstract available. PMID 23130126
- [Background] Alexander KM, Orav J, Singh A, Jacob SA, Menon A, Padera RF, Kijewski MF, Liao R, Di Carli MF, Laubach JP, Falk RH, Dorbala S. Geographic Disparities in Reported US Amyloidosis Mortality From 1979 to 2015: Potential Underdetection of Cardiac Amyloidosis. JAMA Cardiol. 2018 Sep 1;3(9):865-870. doi: 10.1001/jamacardio.2018.2093. PMID 30046835
- [Background] Donnelly JP, Hanna M. Cardiac amyloidosis: An update on diagnosis and treatment. Cleve Clin J Med. 2017 Dec;84(12 Suppl 3):12-26. doi: 10.3949/ccjm.84.s3.02. PMID 29257735
- [Background] Gilstrap LG, Dominici F, Wang Y, El-Sady MS, Singh A, Di Carli MF, Falk RH, Dorbala S. Epidemiology of Cardiac Amyloidosis-Associated Heart Failure Hospitalizations Among Fee-for-Service Medicare Beneficiaries in the United States. Circ Heart Fail. 2019 Jun;12(6):e005407. doi: 10.1161/CIRCHEARTFAILURE.118.005407. Epub 2019 Jun 7. PMID 31170802

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT07314268/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT07314268/ICF_001.pdf